CLINICAL TRIAL: NCT02112994
Title: A Multi-Center, Open-Label Study of Sebelipase Alfa in Patients With Lysosomal Acid Lipase Deficiency
Brief Title: Safety and Efficacy Study of Sebelipase Alfa in Participants With Lysosomal Acid Lipase Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAL-CL06; 2011-004287-30 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-04-14 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: Enzyme Replacement Therapy (ERT); Lysosomal Storage Disease; Late Onset Lysosomal Acid Lipase (LAL) Deficiency; Acid cholesteryl ester hydrolase deficiency, type 2; Acid lipase disease; Cholesterol ester hydrolase deficiency; LAL Deficiency; LIPA Deficiency; Wolman disease; Additional relevant MeSH terms:; Cholesterol Ester Storage Disease; Metabolic Diseases; Lipidoses; Lipid Metabolism, Inborn Errors; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Lysosomal Storage Diseases; Lipid Metabolism Disorders; Infant, Newborn, Diseases
MeSH Terms: conditions — Wolman Disease; Lysosomal Storage Diseases; Cholesterol Ester Storage Disease; Metabolic Diseases; Lipidoses; Lipid Metabolism, Inborn Errors; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Lipid Metabolism Disorders; Infant, Newborn, Diseases | interventions — Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sebelipase Alfa (Experimental): Pediatric and adult participants initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg every week (qw) was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
  Interventions: Drug: Sebelipase Alfa

INTERVENTIONS:
Drug: Sebelipase Alfa — IV infusion of sebelipase alfa
  Other Names: SBC-102

SUMMARY:
This study evaluated the safety and efficacy of sebelipase alfa in a broad population of participants with lysosomal acid lipase deficiency (LAL-D).

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety of intravenous (IV) infusions of sebelipase alfa in a more broad population of LAL-D participants than previously studied. Such participants may have been excluded from enrollment in other studies of LAL-D because of age, disease progression, previous treatment by hematopoietic stem cell or liver transplantation, less common disease manifestations, or disease characteristics that would preclude participation in a placebo-controlled study. This open-label study included infants >8 months, children, and adults. At least 4 participants in the study were to be between the age of 2 and 4 years. Eligible participants received sebelipase alfa at a dose of 1 milligram/kilogram (mg/kg) every other week (qow).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant was >8 months of age at the time of dosing.
2. Confirmation of LAL-D diagnosis as determined by the central laboratory or, for participants with prior hematopoietic stem cell transplant or liver transplant, historical enzyme activity or molecular genetic testing confirming a diagnosis of LAL-D.
3. Participants >8 months but <4 years of age at Screening had at least 1 of the following documented clinical manifestations of LAL-D:

   * Dyslipidemia
   * Elevated transaminases
   * Impaired growth
   * Suspected malabsorption
   * Other clinical manifestation of LAL-D
4. Participants ≥4 years of age at Screening had at least 1 of the following documented clinical manifestations of LAL-D:

   * Evidence of advanced liver disease
   * Histologically confirmed disease recurrence in participants with past liver or hematopoietic transplant
   * Persistent dyslipidemia
   * Suspected malabsorption
   * Other clinical manifestation of LAL-D

Key Exclusion Criteria:

1. Participant had known causes of active liver disease other than LAL-D, which had not been adequately treated.
2. Participant received a hematopoietic stem cell or liver transplant <2 years from the time of dosing.
3. Participant with co-morbidities other than complications due to LAL-D, which were irreversible or associated with a high mortality risk within 6 months or would interfere with study compliance or data interpretation.

Min Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (3):
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Cincinnati, Ohio
- Westmead, Australia
- Brussels, Belgium
- São Paulo, Brazil
- Halifax, Nova Scotia, Canada
- Zagreb, Croatia
- Copenhagen, Denmark
- Freiburg im Breisgau, Germany
- Padua, Italy
- Mexico City, Mexico
- Amsterdam, Netherlands
- Moscow, Russia
- Spain (3):
  - A Coruña
  - Barcelona
  - Madrid
- Balcalı, Turkey (Türkiye)
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Burton BK, Sanchez AC, Kostyleva M, Martins AM, Marulkar S, Abel F, Baric I. Long-Term Sebelipase Alfa Treatment in Children and Adults With Lysosomal Acid Lipase Deficiency. J Pediatr Gastroenterol Nutr. 2022 Jun 1;74(6):757-764. doi: 10.1097/MPG.0000000000003452. Epub 2022 Apr 19. PMID 35442238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 21 study centers were initiated in 15 countries, including Australia, Belgium, Brazil, Canada, Croatia, Denmark, Germany, Italy, Mexico, Netherlands, Russia, Spain, Turkey, United Kingdom (UK), and the United States. Seventeen study centers screened at least 1 participant in all of these countries, except the UK and the Netherlands.
Pre-assignment Details: All participants began treatment with sebelipase alfa at a dose of 1 milligram/kilogram (mg/kg) every other week (qow). Individual participants could escalate/decrease their dose at any time during the study and only at the discretion of the Investigator and in consultation with the Sponsor. All 5 different doses are presented as Milestones below.
Groups:
- 2-<4 Years: This subgroup is part of the full analysis set and includes only participants between the ages of 2 and 4 years old who initiated intravenous (IV) treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg every week (qw) was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
- 4-18 Years: This subgroup is part of the full analysis set and includes only participants between the ages of 4 and 18 years old who initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg qw was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
- >18 Years: This subgroup is part of the full analysis set and includes only participants greater than 18 years old. This subgroup is part of the full analysis set and includes only participants greater than 18 years old who initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg qw was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
Period: Overall Study
Arm/Group | 2-<4 Years | 4-18 Years | >18 Years
Started | 6 | 16 | 9
Received at Least 1 Dose of Study Drug | 6 | 16 | 9
Received 0.35 mg/kg QOW | 0 | 0 | 1
Received 1 mg/kg QOW (All participants started the study at this dose.) | 6 | 16 | 9
Received 1 mg/kg QW | 1 | 1 | 0
Received 3 mg/kg QOW | 3 | 5 | 3
Received 3 mg/kg QW | 2 | 1 | 1
Completed 96-week Treatment Period | 6 | 14 | 8
Completed (Participants who transitioned to commercial product are displayed as having completed the study.) | 6 | 14 | 6
Not Completed | 0 | 2 | 3
Not completed — Progressive Disease | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Liver Transplant | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sebelipase Alfa: Pediatric and adult participants initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg qw was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
Arm/Group | Sebelipase Alfa
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.82 (14.674)
Age, Customized [Count of Participants; unit: Participants]
  2 to <4 years | 6
  4 to 18 years | 16
  >18 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Severe Treatment-emergent Adverse Events (TEAEs)
Description: The number of participants experiencing severe TEAEs is presented for participants who received sebelipase alfa in this open-label study. Adverse events (AEs) information was obtained at each scheduled contact with the participant (or participant's parent or legal guardian). An AE was defined as any untoward medical occurrence that did not require a causal relationship with study drug administration. An AE could have been any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug. Pre-existing conditions that worsened in severity during the study were reported as AEs. A summary of all serious and other non-serious AEs regardless of causality is located in the Reported AE module. Severity assessed using Clinical Data Interchange Standards Consortium Study Data Tabulation Model standard terminology v3.1.1. Data presented only according to age group, not dose of study drug received.
Time Frame: Screening, Week 144
Population: Full Analysis Set: All participants who received at least 1 infusion of sebelipase alfa. The full analysis set was used for analysis of safety and efficacy.
Measure: Count of Participants; unit: Participants
Groups:
- 2-<4 Years: This subgroup is part of the full analysis set and includes only participants between the ages of 2 and 4 years old who initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg qw was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
Arm/Group | 2-<4 Years | 4-18 Years | >18 Years
Number analyzed (Participants) | 6 | 16 | 9
Participants | 1 | 1 | 2

2. Secondary Outcome: Percent Change In Serum Lipids From Baseline To Week 144
Description: The effect of sebelipase alfa on lipid metabolism was evaluated by measuring the change from baseline to Week 144 in 4 serum lipids: low-density lipoprotein cholesterol (LDL-C); high-density lipoprotein cholesterol (HDL-C); non-HDL-C; triglycerides. Blood samples for these clinical laboratory tests were collected at scheduled time points and analyzed by a central laboratory.
Time Frame: Baseline, Week 144
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent Change
Arm/Group | 2-<4 Years | 4-18 Years | >18 Years
Number analyzed (Participants) | 5 | 12 | 2
Percent Change
  LDL-C | -37.5 [-52 to -25] | -29.2 [-59 to 23] | -22.5 [-37 to -8]
  HDL-C | 76.5 [30 to 132] | 24.2 [-4 to 90] | 6.1 [-10 to 22]
  Non-HDL-C | -39.1 [-53 to -29] | -26.7 [-62 to 19] | -22.1 [-33 to -11]
  Triglycerides | -48.3 [-61 to -11] | -15.8 [-74 to 112] | -22.0 [-25 to -19]

3. Secondary Outcome: Participants Testing Positive For Anti-drug Antibodies (ADAs)
Description: The impact of ADAs on the safety and immunogenicity of sebelipase alfa was evaluated by testing for ADAs in participants who received sebelipase alfa in this open-label study. Blood samples for assessment were collected prior to study infusions at Week 2, Week 4, Week 8, Week 12, and every 12 weeks thereafter. Participants testing positive for ADAs were also tested for the presence of neutralizing antibodies that inhibited sebelipase alfa enzyme activity and/or cellular uptake. Any participant experiencing a moderate or severe infusion-associated reaction (IAR) was to have an additional assessment of ADAs at the next study visit (prior to study drug infusion); these participants were to also have serum samples collected at 1 to 2 hours after IAR onset and at the next study visit (prior to study drug infusion) for analysis of serum tryptase. The count of participants who became ADA positive and who tested positive for neutralizing antibodies are presented.
Time Frame: Week 144
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sebelipase Alfa
Number analyzed (Participants) | 31
Participants
  ADA Positive | 2
  Neutralizing Antibodies Positive | 0

4. Secondary Outcome: Percent Change In Body Mass Index (BMI)-For-Age Percentile From Baseline To Week 144 In Pediatric Participants
Description: To evaluate the effects of sebelipase alfa on growth parameters in pediatric participants (≤18 years old) presenting with evidence of growth delay, the percent change in the anthropometric parameter of BMI-for-age percentile from Baseline to Week 144 is reported. Anthropometric parameters were plotted on standard growth curves. When possible, historical data on growth parameters was also incorporated into the analyses. Percentiles and Z-scores for BMI-for-age were determined using standard growth charts appropriate to a participant's age on the date of the assessment: the World Health Organization standard growth chart for participants ≤2 years of age and the Centers for Disease Control standard growth chart for participants >2 years of age.
Time Frame: Baseline, Week 144
Population: Full Analysis Set: All pediatric participants who received at least 1 infusion of sebelipase alfa. The full analysis set was used for analysis of safety and efficacy.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Pediatric Participants: Pediatric participants initiated IV treatment with sebelipase alfa at a dose of 1 mg/kg qow. Participants were considered for a dose adjustment at the discretion of the Investigator and in consultation with the Sponsor. Dose escalation to 3 mg/kg qow was considered if pre-defined dose-escalation criteria were met. If these criteria continued to be met, a subsequent dose escalation to 3 mg/kg qw was considered. Dose decreases as low as 0.35 mg/kg qow were permitted based upon evidence of intolerance to sebelipase alfa treatment. Participants who completed the 96-week treatment period were permitted to continue receiving sebelipase alfa in an expanded treatment period for up to 48 weeks, pending local drug availability and study participation status.
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 17
Percent Change | 26.45 (118.432)

5. Secondary Outcome: Shift In Child-Pugh Status From Baseline To Week 144
Description: In order to evaluate the effects of sebelipase alfa on liver function, the number of participants with a shift in Child-Pugh status from Baseline to Week 144 is reported. The status is based on the Child-Pugh score, which is used in clinical practice to assess prognosis in individuals with chronic liver disease. Laboratory data were used in derivation of the score by summing individual scores (scored 1-3, with 3 indicating most severe) from clinical laboratory test results and physical examinations, including total serum bilirubin, serum albumin, prothrombin time, ascites, and hepatic encephalopathy. The total score was used to determine the Child-Pugh status, reported as Class A (score of 5 or 6), Class B (score of 7 to 9), or Class C (score of 10 to 15). Higher scores and higher categories represented a worse outcome. Data reported as 1 of 2 types of shifts in class: No Change from Baseline; Decline from Baseline.
Time Frame: Baseline, Week 144
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sebelipase Alfa
Number analyzed (Participants) | 18
Participants
  No Change: A to A | 16
  No Change: B to B | 1
  Decline: A to B | 1

ADVERSE EVENTS:
Time Frame: Screening (up to 45 days prior to start of treatment) to Week 144.
Description: All serious and non-serious AE data are displayed by the study drug administered at the time of AE onset.
Groups:
- 0.35 mg/kg QOW: This reporting group is based on the safety set and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 0.35 mg/kg qow.
- 1.0 mg/kg QOW: This reporting group is based on the safety set and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 1.0 mg/kg qow.
- 1.0 mg/kg QW: This reporting group is based on the safety set and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 1.0 mg/kg qw.
- 3.0 mg/kg QOW: This reporting group is based on the safety set and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 3.0 mg/kg qow.
- 3.0 mg/kg QW: This reporting group is based on the safety set and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 3.0 mg/kg qw.
Arm/Group | 0.35 mg/kg QOW | 1.0 mg/kg QOW | 1.0 mg/kg QW | 3.0 mg/kg QOW | 3.0 mg/kg QW
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/31 | 0/2 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 8/31 | 0/2 | 3/11 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 30/31 | 0/2 | 10/11 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.35 mg/kg QOW (N=1) | 1.0 mg/kg QOW (N=31) | 1.0 mg/kg QW (N=2) | 3.0 mg/kg QOW (N=11) | 3.0 mg/kg QW (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Liver transplant (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 0.35 mg/kg QOW (N=1) | 1.0 mg/kg QOW (N=31) | 1.0 mg/kg QW (N=2) | 3.0 mg/kg QOW (N=11) | 3.0 mg/kg QW (N=4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular dilatation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Delayed puberty (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 11 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 12 | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 1
Oral contusion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tongue eruption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 9 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 15 | 0 | 4 | 1
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 2 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 6 | 0 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 13 | 0 | 4 | 3
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Otitis media acute (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 6 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 7 | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 7 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 3 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 3 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 10 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1/3 — Only male participants were exposed to this adverse event.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT02112994/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02112994/SAP_001.pdf